CLINICAL TRIAL: NCT01873352
Title: Evaluate Renal Artery Denervation In Addition to Catheter Ablation To Eliminate Atrial Fibrillation (ERADICATE--AF) Trial
Brief Title: Renal Artery Denervation In Addition to Catheter Ablation To Eliminate Atrial Fibrillation
Acronym: ERADICATE--AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RADCA01
Record Dates: First submitted 2013-06-05; First posted 2013-06-10 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation; Hypertension
MeSH Terms: conditions — Atrial Fibrillation; Hypertension | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CA+RD (Active Comparator): Catheter ablation of atrial fibrillation plus renal sympathetic denervation
  Interventions: Procedure: catheter ablation; Procedure: renal sympathetic denervation
- CA (control) (Active Comparator): Catheter ablation of atrial fibrillation (control group)
  Interventions: Procedure: catheter ablation

INTERVENTIONS:
Procedure: catheter ablation — Patient anesthesia will be administered according to standard EP lab protocol. Arterial and venous access will be achieved through cannulation of the right and/or left femoral arteries and veins as per the usual practice of the EP lab. Full systemic anticoagulation will be instituted as per standard hospital procedures to a target ACT of approximately 300 seconds or greater. Intravascular ultrasound may be used to assist in the positioning of study catheters during the procedure. The AF ablation procedure will be performed using a cryoballoon ablation catheter. Complete pulmonary vein isolation will be the goal of the ablation procedure and PV isolation must be confirmed by a multielectrode mapping catheter within each PV. Pulmonary vein isolation is the only intervention. A cavo-tricuspid isthmus line may be placed in patients with either a history of ECG-determined typical flutter or induced typical flutter during the procedure.
Procedure: renal sympathetic denervation — Right or left femoral artery access. Real-time 3D aorta-renal artery maps constructed with the use of a navigation system and ablation catheter. Mapping and ablation performed after PVI and under identical sedation protocol used for AF ablation. RF delivery of 6 watts to be applied discretely from the first distal main renal artery bifurcation all the way back to the ostium; RF duration of each delivery 1.5 mins; lesions delivered at multiple sites based on multipolar catheter position within renal artery. Use of specifically designed RF delivery system for renal artery denervation is mandatory (RDN). To confirm renal denervation, high-frequency stimulation (HFS) will be applied before the initial and after each RF delivery within the renal artery. Rectangular electrical stimuli will be delivered at the ostium of the targeted renal artery at a frequency of 20 Hz, with an amplitude 15 V and pulse duration of 10 ms for 10 secs.
  Arms: CA+RD

SUMMARY:
The objective of this trial is to determine the role of renal sympathetic denervation in the prevention of atrial fibrillation (AF) recurrence in patients with hypertension for whom a catheter-based AF ablation procedure is planned. Patients will be randomized to either AF catheter ablation (usual therapy) or AF catheter ablation plus renal sympathetic denervation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* History of PAF and plans for a guideline-supported catheter ablation procedure. Paroxysmal AF is defined as AF with duration of 30 secs to 7 days.
* History of significant hypertension (defined as SBP ≥130 mm Hg and/or DBP ≥80 mmHg) and receiving treatment with at least one anti-hypertensive medication
* Renal vasculature accessible as determined by pre-procedural renal MRA
* Willingness to comply with all post-procedural follow-up requirements and to sign informed consent

Exclusion Criteria:

* Inability to undergo AF catheter ablation (e.g., presence of a left atrial thrombus, contraindication to all anticoagulation)
* Prior left atrial ablation for an atrial arrhythmia
* NYHA class IV congestive heart failure
* Pers or longstanding Pers AF (duration > 7 days)
* Renal artery anatomy that is ineligible for treatment
* An estimated glomerular filtration rate (eGFR) < 45mL/min/1.73m2, using the MDRD calculation
* Life expectancy <1 year for any medical condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2013-06-20 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
AAD-free freedom from AF/atrial flutter/atrial tachycardia recurrence at least 30 seconds | 12 months

SECONDARY OUTCOMES:
Freedom from AF recurrence (not-including the pre-defined 3 month blanking period) despite taking AADs | 12 months
Blood pressure control between the two groups as compared to baseline | 6 months
Blood pressure control between the two groups as compared to baseline | 12 months
Differences in measures of LV hypertrophy/compliance (LV wall thickness, mitral inflow parameters) and LA size | 12 months
Procedure adverse events | 12 months
Major adverse cardiac events (defined as a composite of: death, stroke, CHF hospitalization, clinically diagnosed thromboembolic events other than stroke and hemorrhage requiring transfusion) | 12 months
Serious adverse events throughout follow-up | 12 months
Total number of anti-hypertensive medications at study end, compared between the two treatment arms | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Pokushalov, MD, PhD, Principal Investigator — State Research Institute of Circulation Pathology; Jonathan S. Steinberg, MD, Principal Investigator — University of Rochester
Locations (2):
- Jonathan S. Steinberg, Short Hills, New Jersey, United States
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- [Derived] Steinberg JS, Shabanov V, Ponomarev D, Losik D, Ivanickiy E, Kropotkin E, Polyakov K, Ptaszynski P, Keweloh B, Yao CJ, Pokushalov EA, Romanov AB. Effect of Renal Denervation and Catheter Ablation vs Catheter Ablation Alone on Atrial Fibrillation Recurrence Among Patients With Paroxysmal Atrial Fibrillation and Hypertension: The ERADICATE-AF Randomized Clinical Trial. JAMA. 2020 Jan 21;323(3):248-255. doi: 10.1001/jama.2019.21187. PMID 31961420
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru